CLINICAL TRIAL: NCT03653234
Title: TV-based Assistive Integrated Service to Support European Adults Living With Mild Dementia or Mild Cognitive Impariment
Brief Title: TV-based Service to Support People Living With Mild Dementia or Mild Cognitive Impariment
Acronym: TV-AssistDem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Îngrijiri la domiciliu, Romania (Unknown); Consiglio Nazionale delle Ricerche, Italy (Unknown); Institut multidisciplinaire de science de données, Italy (Unknown); Asociación de Familiares de Personas con Alzheimer y otras Demencias de Málaga, Spain (Unknown); Smart Health TV Solution, Spain (Unknown); Istituto di Scienze e Tecnologie della Cognizione, Switzerland (Unknown); MEDEA, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TV-AssistDem (AAL-2016-024)
Record Dates: First submitted 2018-07-11; First posted 2018-08-31 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2020-05

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
Keywords: active and assisted living; assistive technology; telecare; remote consultations; informal caregivers; quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TV-based Assistive Integrated Service (Experimental): Participants assigned to the intervention group will have access to TV-AssistDem and participate in clinical visits every 6 months.
  Interventions: Device: TV-based Assistive Integrated Service
- Control (No Intervention): Participants assigned to the intervention group will NOT have access to TV-AssistDem and will participate in clinical visits every 6 months

INTERVENTIONS:
Device: TV-based Assistive Integrated Service — TV-AssistDem is an interactive platform which has been adapted specifically for people with MCI and mild dementia through a structured process. The application is intended to be used daily at home, mainly by the participants themselves, with the help of their informal caregivers. The device consists of an Android software and hardware TV (a Digital TV STB with Android technology).
  The core services of the platform are: 1) Calendar and reminders, 2) Health tracking and data transmission and 3) Videoconference; service-oriented applications are: 4) Cognitive stimulation (Stimulus© software); 5) Reminiscences; and 6) Patient and caregiver advice.
  Arms: TV-based Assistive Integrated Service

SUMMARY:
This multicentre randomized controlled trial aims to evaluate the effects of an intervention consisting of a TV-based Assistive Integrated Service developed to improve the quality of life in older people with mild cognitive impairment or mild dementia (PMCI/MD) and their informal caregivers. This study is a collaboration between four European countries (Spain, Romania, Italy and Switzerland) and the clinical trials will be conducted in two of these countries (Spain and Romania) In total 240 dyads, consisting of a person with mild cognitive impairment or mild dementia and their informal caregiver will be recruited for this study. Participant dyads will be randomized in a 1:1 ratio in two parallel groups: to receive either usual care from primary or specialized providers (control group) or to receive usual care plus access to a device with the Tv-AssistDem platform (intervention group).

Participants in the trial will be assessed for a period of 12 months. After the baseline visit, all participants will have follow-up visits every 6 months together with a checkup of the PMCI/MD capacity to remain in the study. In the follow up visits, investigators will assess the PMCI/MD quality of life, caregiver's quality of life and burden, patient treatment adherence, patient functional status and service utilization. A user-behaviour analysis and usability evaluation will also be performed.

DETAILED DESCRIPTION:
TV-AssistDem is an interactive platform which has been designed and developed adapting the functionalities and content to best fit PMCI/MD, in a process involving the structured participation of PMCI/MD, their informal caregivers, and clinicians.

QUALITY ASSURANCE PLAN. The researchers will review and report the process during the trial covering participant enrolment, consent, eligibility and allocation to trial groups, policies to protect participants, including reporting of harm and completeness, accuracy and timeliness of data collection.

STANDARD OPERATING PROCEDURES. Participants will be recruited over a period of three months by physicians (primary care, psychiatry, neurology, and geriatrics), neuropsychologists and dementia and mental health nurses. Participants will not receive financial reimbursement for taking part in this trial. Participants will be identified from people with self- perceived cognitive impairment or caregiver´s perception of cognitive impairment that has been present for more than six months and who meet all the study eligibility criteria (listed in section Eligibility). The Mini-Mental State Examination (MMSE) and Geriatric Depression Scale (GDS-15) will be used to screen PMCI/MD at recruitment. Participants can be under primary care services as well as secondary care services. Participants will also be identified from patient databases such as those integrated in the network.

DATA DICTIONARY. All variables collected in this study are listed and described in an electronic case report form, with associated guidelines, to ensure consistency in all gathered data. The following data will be collected in this trial:

* Sociodemographical data.
* Medical history - PMCI/MD only.
* Quality of Life-Alzheimer's Disease Scale (QoL-AD Scale) (1-3).
* European Quality of Life 5 Dimensions 5 Levels (EuroQoL-5D-5L) (4,5).
* Zarit Burden Interview (ZBI-12) (6,7).
* Treatment adherence: Pill/dose count (8-10) and Morisky-Green Test (11).
* Functional decline: Lawton - Brody Instrumental Activities Of Daily Living Scale (IADL) (12).
* Service Utilisation: Client Service Receipt Inventory (CSRI) (13,14).
* Data from the TV-AssistDem application focusing on User-behaviour and usage of core services.
* Usability Evaluation: System Usability Scale (SUS) (15,16).

SAMPLE SIZE ASSESSMENT. The main outcome measure is the total score of the QoL-AD, which ranges from 13 to 52. According to recent studies (17,18) , the standard deviation of the total score of the QoL-AD is 7. For a minimum important clinical difference of 2.77 on the total QoL-AD score, with a standard deviation of 7, the effect size is 0.39.

To compare two groups (Intervention and Control) using a two- sample, two-sided t-test with a 5% statistical significance level, the minimum number of evaluable PMCI/MDs required in each group is 100 (200 overall), to give a power of 80%. If there would be a drop-out rate of 20% of the PMCI/MDs then the number of PMCI/MDs registered on the study would need to be 120 in each group (240 overall).

STATISTICS ANALYSIS PLAN. The flow of individuals will be shown schematically with counts and percentages in a CONSORT diagram. The analysis will be made following an intention-to-treat procedure. All variables collected will be summarized by group and by site at baseline and at final follow-up. Statistics considered for presentation for continuous measures in summary tables will be the mean, minima and maxima, and standard deviation, and if the criteria of normality are not met, the median and the first and third quartiles. Categorical variables will be summarized using counts and percentages. The baseline variables of the experimental group and the control group will be compared using the Chi-Square test for categorical variables and analysis of covariance for continuous variables.

For the primary outcome, a Linear Mixed Model analyses will be carried out as this approach is optimal to include subjects with missing data. First, an unadjusted analysis will be carried out and secondarily, in case that potentially confusing factors differ between the experimental group and the control group, despite the randomization, a supplementary multivariate analysis will be carried out. For secondary outcomes a Linear Mixed Model and Generalized Mixed Model analysis will be used for continuous and categorical variables respectively. Analysis will be two-tailed and alpha level set at 0.05.

ECONOMIC ANALYSIS. A cost-effectiveness and/or cost-utility analysis from a Health Service perspective (financer perspective) will be performed. The time horizon is two years and will include only direct costs. This refers to direct health costs (medication and healthcare use of services including outpatient and emergencies visits and hospital admissions). The Quality-Adjusted Life Years (QALYs) will be calculated to estimate the benefit calculating the utility improvement measure by EuroQoL-5D-5L.

USER-BEHAVIOUR ANALYSIS AND USABILITY EVALUATION. Data on various platform usage variables will be collected for the intervention group. Regression analysis will be used to assess the relationship between the primary and secondary outcome variables and the usage variables in order to indicate which aspects of the computer platform use most affect the outcomes. The results of the usability tests will be analyzed using statistical methods to quantify the error rate, effectiveness and learning curve of the TV-AssistDem platform.

PLAN FOR MISSING DATA. Each researcher is responsible for ensuring that any missing data will be reported as missing in the study database. Procedures can sometimes be considered when using statistical methods that fail in the presence of any missing values, or when in the case of multiple-predictor statistical models all the data for an individual would be omitted because of a missing value in one of the predictors. For analyses involving multiple regression analysis, a multiple imputation approach will be considered and used if statistically sound, depending on the proportion and pattern of missing values.

METHODS TO ENSURE VALIDITY AND QUALITY OF DATA. Accurate and reliable data collection will be assured by verification and cross-check of the case report form (CRF) against the researcher´s records (source document verification). Source document verification will be conducted for 5% of data in subjects. A comprehensive validation check program utilizing front-end checks in the CRF will verify these data. Discrepancies and queries will be generated accordingly in the CRF for online resolution by the researcher at the site. In addition, the CRF data will be reviewed on an ongoing basis for medical and scientific plausibility.

ELIGIBILITY:
Inclusion Criteria:

* Participants score 23-27 points on Mini-Mental State Examination (MMSE).
* Self-perceived cognitive impairment or caregiver´s perception of cognitive impairment that has been present for more than six months.
* Participants +60 years of age.
* Participants live independently.
* Participants have an informal caregiver.
* Participants who take prescribed medication are in charge of their own medication use.
* Participant with pharmacological treatment for a chronic conditions during study period.
* The place where the participant is normally resident has enough wireless or phone network connectivity to enable them to use Tv-AssistDem platform on a daily basis.
* Participants agree to be part of the study by giving signed written consent.

Exclusion Criteria:

* Participants have a terminal illness with <3 years expected survival.
* Participants score above 11 on the Geriatric Depression Scale (GDS-15).
* Participants have specific conditions reducing their physical ability to use the application to a point that makes their participation in the project impossible (the nature of the conditions will be recorded in such cases).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of life in people with mild cognitive impairment or mild dementia at 6 and 12 months. | At baseline and then at 6 and 12 months.
  Quality of Life-Alzheimer's Disease Scale (QoL-AD Scale) (1-3) is an instrument specifically designed to measure quality of life in people with dementia from the perspective of both the patient and the informal caregiver. It is a 13-item measure, which includes assessments of the person´s relationships with friends and family, financial situation, physical condition, mood, memory and an overall assessment of life quality. Response options are 4-point multiple choice options (1 = poor, 2= fair, 3= good, 4 = excellent). Scale scores range from 13 to 52, with higher scores indicating greater quality of life.
  PMCI/MD may lose cognitive function during the study to the extent that they are unable to complete the assessments themselves. For this reason, informal caregivers will also complete the QoL-AD, in parallel and on behalf of the PMCI/MD, from the start of the study.

SECONDARY OUTCOMES:
Change from baseline quality of life in informal caregivers at 6 and 12 months. | At baseline and then at 6 and 12 months.
  European Quality of Life 5 Dimensions 5 Levels (EuroQoL-5D-5L) (4,5) is a standardized generic instrument consisting of a descriptive system and a visual analogue scale (VAS). The descriptive system comprises 5 dimensions covering mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A 1-digit number expresses the level selected for that dimension. The digits can be combined into a 5-digit number that describes the patient's health state. The VAS records the patient's self-rated health on a vertical scale, where the endpoints are 'The best health you can imagine' and 'The worst health you can imagine'.
  EuroQoL-5D-5L has been shown to correlate well with QoL-AD, indicating that using both measures side-by-side is compatible. Both will be completed by the patient and caregiver.
Change from baseline burden in informal caregivers at 6 and 12 months. | At baseline and then at 6 and 12 months.
  Zarit Burden Interview (ZBI-12) (6,7) is a 12-item scale with each answer chosen from a 5-point Likert scale (Nearly always=4, Quite frequently=3, Sometimes=2, Rarely=1, Never=0). It is a shortened version of the original scale, was developed specifically for informal caregivers of PMCI/MD and covers issues such as caregiver stress and the degree to which caring is affecting their health and social life. Total score range 0 to 48 (0-10= no to mild burden, 10-20= mild to moderate burden >20= high burden).
Change from baseline treatment adherence in people with mild cognitive impairment or mild dementia at 6 and 12 months. | At baseline and then at 6 and 12 months.
  The dose/pill count (8-10) is the number of pills or doses taken divided by the prescribed ones, multiplied by 100 (expressed as a percentage). A good adherence is considered when the result of counting is between 80% (a twenty percent of doses/pills missed) and 110% (the patient takes ten percent more doses/pills) of dose/pill prescribed.
Change from baseline treatment compliance in people with mild cognitive impairment or mild dementia at 6 and 12 months. | At baseline and then at 6 and 12 months.
  The Morisky Green Test (11) consists of 4 contrast questions with dichotomous yes/no responses, reflecting the patient's behaviour regarding compliance. They are intended to assess whether the patient adopts correct attitudes regarding treatment for their disease; it is assumed that if the attitudes are incorrect the patient is non-compliant.
Change from baseline functional decline in people with mild cognitive impairment or mild dementia at 6 and 12 months. | At baseline and then at 6 and 12 months.
  Lawton Instrumental Activities of Daily Living (IADL) (12) is an interview format scale of 8-items covering instrumental activities, which are required for independent living: ability to use telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsability for own medications and ability to handle finances. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change from baseline healthcare costs at 12 months | At baseline and then at 12 months
  The Client Service Receipt Inventory (CSRI) (13,14) is an internationally used method for gathering data on service utilization and other domains relevant for economic analysis of mental health care. It has five sections: background client information, accommodation and living situation, employment history, earnings and benefits, a record of services usually used and information about informal caregiver support. The sections assessed will be consultations, admissions and visits in the last year, grouped into subsections according to hospital, specialist, primary or home care. Treatment related to hospital admissions or illness exacerbation will also be assessed.
  It´s adaptability ensures it is compatible with the research aims, context, participants' likely circumstances, and the quantity and precision of information required

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Mayoral Cleries, Principal Investigator — Instituto de Investigación Biomédica de Malaga (IBIMA)-Fundacion FIMABIS
Locations (2):
- Îngrijiri La Domiciliu, Brasov, Romania
- Instituto de Investigacion Biomedica de Malaga-IBIMA, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thorgrimsen L, Selwood A, Spector A, Royan L, de Madariaga Lopez M, Woods RT, Orrell M. Whose quality of life is it anyway? The validity and reliability of the Quality of Life-Alzheimer's Disease (QoL-AD) scale. Alzheimer Dis Assoc Disord. 2003 Oct-Dec;17(4):201-8. doi: 10.1097/00002093-200310000-00002. PMID 14657783
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Logsdon, R.G., Gibbons, L.E., McCurry, S.M., & Teri L. Quality of life in Alzheimer's disease: Patient and caregiver reports. J Ment Heal Aging. 1999;5(1):21-32.
- [Background] Gomez-Gallego M, Gomez-Amor J, Gomez-Garcia J. [Validation of the Spanish version of the QoL-AD Scale in alzheimer disease patients, their carers, and health professionals]. Neurologia. 2012 Jan;27(1):4-10. doi: 10.1016/j.nrl.2011.03.006. Epub 2011 May 12. Spanish. PMID 21570161
- [Background] Devlin NJ, Krabbe PF. The development of new research methods for the valuation of EQ-5D-5L. Eur J Health Econ. 2013 Jul;14 Suppl 1(Suppl 1):S1-3. doi: 10.1007/s10198-013-0502-3. No abstract available. PMID 23900659
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Sackett DL, Haynes RB, Gibson ES, Hackett BC, Taylor DW, Roberts RS, Johnson AL. Randomised clinical trial of strategies for improving medication compliance in primary hypertension. Lancet. 1975 May 31;1(7918):1205-7. doi: 10.1016/s0140-6736(75)92192-3. PMID 48832
- [Background] Hansen RA, Kim MM, Song L, Tu W, Wu J, Murray MD. Comparison of methods to assess medication adherence and classify nonadherence. Ann Pharmacother. 2009 Mar;43(3):413-22. doi: 10.1345/aph.1L496. Epub 2009 Mar 3. PMID 19261962
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Beecham J, Knapp M. 12 Costing psychiatric interventions. In: G. Thornicroft, editor. Measuring Mental Health Needs. 2a. 2001. p. 200-24.
- [Background] Brooke J. SUS : A Retrospective. J Usability Stud. 2013;8(2):29-40.
- [Background] Bangor A, Kortum P, Miller J. Determining what individual SUS scores mean: Adding an adjective rating scale. J usability Stud. 2009;4(3):114-23.
- [Background] Goeman D, Comans T, Enticott JC, Renehan E, Beattie E, Kurrle S, Koch S. Evaluating the Efficacy of the "Support for Life" Program for People with Dementia and Their Families and Carers' to Enable Them to Live Well: A Protocol for a Cluster Stepped Wedge Randomized Controlled Trial. Front Public Health. 2016 Oct 31;4:245. doi: 10.3389/fpubh.2016.00245. eCollection 2016. PMID 27843893
- [Background] Woods RT, Orrell M, Bruce E, Edwards RT, Hoare Z, Hounsome B, Keady J, Moniz-Cook E, Orgeta V, Rees J, Russell I. REMCARE: Pragmatic Multi-Centre Randomised Trial of Reminiscence Groups for People with Dementia and their Family Carers: Effectiveness and Economic Analysis. PLoS One. 2016 Apr 19;11(4):e0152843. doi: 10.1371/journal.pone.0152843. eCollection 2016. PMID 27093052
- [Derived] Goodman-Casanova JM, Dura-Perez E, Guzman-Parra J, Cuesta-Vargas A, Mayoral-Cleries F. Telehealth Home Support During COVID-19 Confinement for Community-Dwelling Older Adults With Mild Cognitive Impairment or Mild Dementia: Survey Study. J Med Internet Res. 2020 May 22;22(5):e19434. doi: 10.2196/19434. PMID 32401215
- [Derived] Goodman-Casanova JM, Guzman-Parra J, Guerrero G, Vera E, Barnestein-Fonseca P, Cortellessa G, Fracasso F, Umbrico A, Cesta A, Toma D, Boghiu F, Dewarrat R, Triantafyllidou V, Tamburini E, Dionisio P, Mayoral F. TV-based assistive integrated service to support European adults living with mild dementia or mild cognitive impairment (TV-AssistDem): study protocol for a multicentre randomized controlled trial. BMC Geriatr. 2019 Sep 6;19(1):247. doi: 10.1186/s12877-019-1267-z. PMID 31492113